CLINICAL TRIAL: NCT04754100
Title: A Phase 1, Open-Label Study of the Safety, Tolerability, and Preliminary Clinical Activity of Allogeneic Invariant Natural Killer T (iNKT) Cells (agenT-797) in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: agenT-797 in Participants With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MiNK Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1305
Record Dates: First submitted 2021-02-03; First posted 2021-02-15 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Multiple myeloma; Immunotherapy; iNKT cells
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogeneic iNKT Cells (Experimental): 3+3 Dose escalation of agenT-797 will be administered by intravenous infusion every 2 weeks (each cycle is 14 days [2 weeks]).
  Interventions: Drug: agenT-797

INTERVENTIONS:
Drug: agenT-797 — agenT-797 is an off-the-shelf cell therapy consisting of ≥ 95% allogeneic human unmodified iNKT cells isolated from 1 healthy donor mononuclear cell apheresis unit and expanded ex vivo.

SUMMARY:
This is a Phase 1, open-label study to explore the safety, tolerability, and preliminary clinical activity of agenT-797, an unmodified, allogeneic iNKT cell therapy, in participants with relapsed or refractory multiple myeloma, as well as to define the recommended Phase 2 dose.

ELIGIBILITY:
Key Inclusion Criteria:

1. Relapsed/Refractory Multiple Myeloma

   1. Confirmed diagnosis and evidence of progressive disease or clinical relapse as defined by International Myeloma Working Group criteria and following prior therapy for multiple myeloma (MM)
   2. Relapsed or refractory MM requiring current treatment
   3. Previously failed ≥ 3 prior regimens (after at least 2 cycles of medication per regimen) and included at least 1 immunomodulatory drug, 1 proteasome inhibitor, and an anti-CD38 antibody agent
   4. Participants must have measurable disease as defined by at least 1 of the following:

      * Serum M-protein ≥ 0.5 grams/deciliter (dL) by serum protein electrophoresis or for immunoglobulin A (IgA) myeloma, by quantitative IgA; or
      * Urinary M-protein excretion at least 200 milligrams (mg)/24 hours; or
      * Serum free light chain whereby the involved light chain measures ≥ 10 mg/dL and with an abnormal ratio
2. Estimated life expectancy ≥ 3 months
3. No other medical, surgical, or psychiatric condition (including active substance abuse) that would interfere with compliance to the protocol, as determined by the principal investigator

Key Exclusion Criteria:

1. Concurrent invasive malignancy
2. Participants who had an allogeneic stem cell transplantation and are still on immunosuppressive medications or corticosteroids above physiological dose within 4 weeks before agenT-797
3. Prior radiotherapy within 2 weeks of start of study treatment
4. Prior systemic cytotoxic chemotherapy, biological therapy, or major surgery within 3 weeks prior to dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number Of Participants With Treatment-related Adverse Events | Baseline through Day 28 post cell infusion
  This will be determined by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0.
Number Of Dose-limiting Toxicities | Baseline through Day 14 post cell infusion

SECONDARY OUTCOMES:
Persistence Of agenT-797 In Peripheral Blood | Baseline/Day 1 (pre-infusion, 5 minutes, 0.25, 0,5, 1, 2, and 4 hours post cell infusion), Days 2, 3, 5, 8, 15, 22, and 29, Weeks 6, 8, and 12, and Months 6, 9, and 12
Overall Response Rate (ORR) | End of study visit (up to 12 months)
Duration Of Response (DOR) | End of study visit (up to 12 months)
Duration Of Clinical Benefit | End of study visit (up to 12 months)
Time To Response (TTR) | End of study visit (up to 12 months)
Measurement Of Serum Alloantibodies To Major Histocompatibility Complex Class I And II | Baseline/Day 1 (pre-infusion), Day 22, Week 6, and end of study visit (up to 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MiNK Therapeutics
Locations (3):
- United States (3):
  - Norton Cancer Institute - St. Matthews - Medical Oncology/Hematology Candida, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Cincinnati Cancer Center, Cincinnati, Ohio